CLINICAL TRIAL: NCT07407192
Title: Toxicity Outcomes of Simultaneous Integrated Boost as Part of Adjuvant Radiotherapy in Breast Cancer Patients After Breast-Conserving Surgery
Brief Title: Toxicity Outcomes of Simultaneous Integrated Boost in Adjuvant Breast Radiotherapy Acronym
Acronym: SIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OI-BREAST-SIB-2019; ERIDEK-0045/2019 (Other: Ethics Committee, Institute of Oncology Ljubljana)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with breast cancer after breast-conserving surgery receive adjuvant radiotherapy with a simultaneous integrated boost (SIB) to the tumor bed. Acute and late toxicity outcomes are prospectively recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Radiotherapy With Simultaneous Integrated Boost (SIB) (Experimental): Breast cancer patients treated with breast-conserving surgery receive adjuvant radiotherapy to the whole breast with a simultaneous integrated boost (SIB) to the tumor bed, using either standard fractionation or hypofractionation. Acute and late toxicity outcomes are prospectively recorded.
  Interventions: Radiation: Adjuvant Breast Radiotherapy With Simultaneous Integrated Boost (SIB)

INTERVENTIONS:
Radiation: Adjuvant Breast Radiotherapy With Simultaneous Integrated Boost (SIB) — Adjuvant whole-breast radiotherapy after breast-conserving surgery with a simultaneous integrated boost (SIB) dose delivered to the tumor bed during the same treatment sessions. Treatment is delivered using either standard fractionation or hypofractionation, according to institutional protocol.

SUMMARY:
This prospective study systematically evaluates toxicity outcomes in breast cancer patients treated with adjuvant radiotherapy using the simultaneous integrated boost (SIB) technique after breast-conserving surgery. The aim is to monitor acute and late treatment-related side effects during implementation of this radiotherapy approach and to compare institutional toxicity outcomes with published data in the literature.

DETAILED DESCRIPTION:
Breast cancer patients undergoing breast-conserving surgery are treated with adjuvant radiotherapy using either standard fractionation or hypofractionation combined with a simultaneous integrated boost (SIB) to the tumor bed. This prospective study includes systematic collection and grading of acute and late radiation-related toxicity outcomes in order to evaluate the safety of the implemented protocol and to assess whether toxicity rates are comparable to those reported in published clinical studies. The results will support optimization and quality assurance of the radiotherapy technique in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Female patients with histologically confirmed breast cancer

Status post breast-conserving surgery (lumpectomy)

Planned adjuvant whole-breast radiotherapy with simultaneous integrated boost (SIB) to the tumor bed

Age ≥ 18 years

Ability to provide informed consent

Exclusion Criteria:

Prior radiotherapy to the breast or thoracic region

Mastectomy (no breast-conserving surgery)

Pregnancy or breastfeeding

Inability to complete planned radiotherapy or follow-up assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Acute Radiation Toxicity (CTCAE) | From start of radiotherapy up to 3 months after completion of radiotherapy
  Incidence and severity of acute radiotherapy-related toxicity assessed during treatment and shortly after completion, graded according to Common Terminology Criteria for Adverse Events (CTCAE).
Acute Radiation Toxicity (CTCAE) | From start of radiotherapy up to 3 months after completion of radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No